CLINICAL TRIAL: NCT05730699
Title: An Open-Label Study of the Efficacy and Safety of Divozilimab in Patients With Neuromyelitis Optica Spectrum Disorders
Brief Title: Efficacy and Safety of Divozilimab in Patients With Neuromyelitis Optica Spectrum Disorders (AQUARELLE)
Acronym: AQUARELLE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCD-132-6
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Neuromyelitis Optica Spectrum Disorders
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCD-132 (divozilimab) (Experimental): Intravenous infusion of BCD-132 every 24 weeks
  Interventions: Biological: divozilimab

INTERVENTIONS:
Biological: divozilimab — anti-CD20 monoclonal antibody

SUMMARY:
The goal of this clinical trial is to study the efficacy and safety of BCD-132 (divozilimab) in subjects with neuromyelitis optica spectrum disorders (NMOSD).

DETAILED DESCRIPTION:
BCD-132-6/AQUARELLE is an open-label phase 3 clinical study in subjects with NMOSD. Approximately 105 subjects will be enrolled.

The study consists of a screening period, a treatment period and a follow-up period. During treatment period, the subjects will receive the investigational product divozilimab.

The duration of participation for each subject will be approximately 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* NMOSD diagnosed based on the 2015 NMOSD International Consensus Diagnostic Criteria
* Documented evidence of at least 1 relapse within 12 months before signing the informed consent form, or 2 relapses within 24 months before signing the informed consent form
* A total EDSS score of ≤ 7
* Presence of IgG antibodies to the Varicella Zoster virus at screening
* A CD19+ cell proportion of ≥ 1 % of the total lymphocyte count in patients exposed to other anti-B-cell therapies more than 6 months before signing the informed consent form

Exclusion Criteria:

* A relapse occurring less than 30 days before signing the informed consent form or at screening (patients may be re-screened)
* Intrathecal oligoclonal or monoclonal IgG production (in patients who are anti-AQP4 seronegative)
* Other nervous system disorders (including multiple sclerosis) that can mask or affect the assessment of NMOSD symptoms
* History of other autoimmune diseases requiring immunosuppressive therapy
* Prior exposure to: alemtuzumab, total lymphatic irradiation, bone marrow transplantation; anti-B-cell therapy drugs, abatacept, satralizumab within 6 months prior to signing the informed consent form; mitoxantrone, cyclophosphamide, methotrexate, cyclosporine A, tacrolimus, eculizumab, tocilizumab, natalizumab, interferon beta, glatiramer acetate, fingolimod, teriflunomide, dimethyl fumarate within 3 months before signing the informed consent form; immunoglobulin products within 30 days before signing the informed consent form; transfusion of blood or blood components within 30 days before signing the informed consent form; systemic corticosteroids at the time of signing the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Adjudicated annualized relapse rate [Week 24] | Week 24
  Adjudicated annualized relapse rate

SECONDARY OUTCOMES:
Time to the first adjudicated relapse | Week 100
  Time to the first adjudicated relapse is defined as the time from the date of randomization in the study to the date of the onset of symptoms of the adjudicated relapse. Each relapse will be adjudicated by an independent neurological commission
Adjudicated annualized relapse rate | Week 52, 100
  Adjudicated annualized relapse rate
Proportion of subjects without adjudicated relapses | Weeks 24, 52, 100
  Proportion of subjects without adjudicated relapses at week 24, 52, 100
Change in the Expanded Disability Status Scale (EDSS) score | Week 24, 52, 100
  Change in the Expanded Disability Status Scale (EDSS) at week 24, 52, 100 relative to baseline.The EDSS ranges from 0 to 10. An increase in EDSS values corresponds to a worsening disability.
Proportion of subjects with confirmed increase in disability | Weeks 24, 26, 48, 52, 100
  Confirmed increase in disability is defined as an increase in the EDSS score (not related to a previous relapse and assuming there is no relapse at assessment) compared to Day 1 (baseline) by at least 1.5 in subjects with a baseline score of 0; by at least 1.0 in subjects with a baseline score of > 0 and ≤ 5.5; and by at least 0.5 in subjects with a baseline score of ≥ 6.0 persisting for ≥ 3 months
Vision acuity change | Week 24, 52, 100
  Vision acuity change at Week 24, 52, 100 relative to baseline
Change in the Timed 25-Foot (7.62 m) Walk (T25-FW) test | Up to Week 100
  Change in the Timed 25-Foot (7.62 m) Walk (T25-FW) test over time compared to baseline.
  T25-FW test is a way to quantify lower limb functions. The subject standing at one end of a clearly marked 25-foot (7.62-meter) course is asked to walk the distance as quickly but as safely as possible. After the first attempt, the subject is asked to walk the same distance again. The results (time in seconds) of both attempts are recorded.
Changes in the severity of pain using a Numeric Rating Scale | Week 4, 24, 52, 100
  Changes in the severity of pain at Week 4, 24, 52, 100 relative to baseline. The Numerical Rating Scale (NRS) will be used to assess the intensity of the subject's pain. NRS consists of consecutive numbers from 0 to 10, where 0 is no pain and 10 is the most severe pain that can be imagined.
Change in the quality of life using a SF-36 | Week 24, 52, 100
  Change in the quality of life parameters using a SF-36 questionnaire at week 24, 52, 100 relative to baseline. SF-36 (Short Form-36) questionnaire includes a total of 36 questions.
CUA | Week 24
  CUA (Cumulative Total Active) - • Cumulative number of new Gd-enhancing T1-weighted lesions and new T2-weighted lesions or enlarging T2-weighted lesions without double counting

CONTACTS AND LOCATIONS:
Locations (19):
- Russia (19):
  - Llc "Profimed", Barnaul
  - Municipal Autonomous Healthcare Institution of the Order of the Red Banner of Labor "City Clinical Hospital No.1", Chelyabinsk
  - Regional Clinical Hospital No.3, Chelyabinsk
  - Kuzbass Clinical Hospital named after S.V. Belyaev, Kemerovo
  - Khanty-Mansiysk autonomous district - Ugra "The district clinical hospital", Khanty-Mansiysk
  - Center for Cardiology and Neurology, Kirov
  - Regional Clinical Hospital № 1 named after Professor S. V. Ochapovsky, Krasnodar
  - Moscow Regional Clinical Research Institute named after M.F. Vladimirsky (MONIKI), Moscow
  - LLC "Medis", Nizhny Novgorod
  - Semashko Regional Clinical Hospital, Nizhny Novgorod
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Pyatigorsk City Clinical Hospital No.2, Pyatigorsk
  - Federal State Budgetary Educational Institution of Higher Education "Rostov State Medical University", Rostov-on-Don
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Seredavin Regional Clinical Hospital, Samara
  - Republican Clinical Hospital No.4, Saransk
  - Siberian State Medical University, Tomsk
  - Medical and Sanitary Unit "Neftyanik", Tyumen
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk